CLINICAL TRIAL: NCT01180075
Title: Tenofovir, Emtricitabine, Efavirenz and Atazanavir Pharmacokinetics in the Aging HIV-Infected Population
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Julie Dumond, PharmD, Assistant Professor, University of North Carolina, Chapel Hill
Other Study IDs: 09-2120; 1K23AI093156-01A1 (NIH)
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Atazanavir Sulfate; Ritonavir; Phlebotomy

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for determining drug concentrations and for future genetic testing of drug metabolizing enzymes and transporters will be stored for up to 5 years.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- TDF/FTC/EFV Intensive Sampling-Group A: Patients receiving TDF/FTC/EFV who undergo intensive pharmacokinetic sampling over 24 hours
  Interventions: Drug: tenofovir/emtricitabine/efavirenz (TDF/FTC/EFV); Procedure: Phlebotomy
- TDF/FTC/ATV/r Intensive Sampling Group A: Patients receiving TDF/FTC/ATV/r who undergo intensive pharmacokinetic sampling over 24 hours
  Interventions: Drug: tenofovir/emtricitabine (TDF/FTC); Drug: Atazanavir (ATV); Drug: Ritonavir; Procedure: Phlebotomy
- TDF/FTC/EFV Sparse Sampling Group B: Patients receiving TDF/FTC/EFV who undergo sparse pharmacokinetic sampling on 1 or 2 visits depending on subject's availability
  Interventions: Drug: tenofovir/emtricitabine/efavirenz (TDF/FTC/EFV); Procedure: Phlebotomy
- TDF/FTC/ATV/r Sparse Sampling Group B: Patients receiving TDF/FTC/ATV/r who undergo sparse pharmacokinetic sampling on 1 or 2 visits depending on subject's availability
  Interventions: Drug: tenofovir/emtricitabine (TDF/FTC); Drug: Atazanavir (ATV); Drug: Ritonavir; Procedure: Phlebotomy

INTERVENTIONS:
Drug: tenofovir/emtricitabine/efavirenz (TDF/FTC/EFV) — Patients receiving this drug for clinical care at standard dosages will be enrolled.
  Other Names: Atripla
  Groups: TDF/FTC/EFV Intensive Sampling-Group A; TDF/FTC/EFV Sparse Sampling Group B
Drug: tenofovir/emtricitabine (TDF/FTC) — Patients receiving this drug for clinical care at standard dosages will be enrolled.
  Other Names: Truvada
  Groups: TDF/FTC/ATV/r Intensive Sampling Group A; TDF/FTC/ATV/r Sparse Sampling Group B
Drug: Atazanavir (ATV) — Patients receiving this drug for clinical care at 300mg with 100mg ritonavir daily will be enrolled.
  Other Names: Reyataz
  Groups: TDF/FTC/ATV/r Intensive Sampling Group A; TDF/FTC/ATV/r Sparse Sampling Group B
Drug: Ritonavir — Patients receiving this drug for clinical care at 100mg daily with 300mg atazanavir will be enrolled.
  Other Names: Norvir
  Groups: TDF/FTC/ATV/r Intensive Sampling Group A; TDF/FTC/ATV/r Sparse Sampling Group B
Procedure: Phlebotomy — Multiple blood draws will be performed in the study, and vary depending on the group.

SUMMARY:
Purpose: To see how growing older changes the amount of HIV drugs in the blood of HIV-infected men and women. Many changes happen in the body as it ages that may affect the way drugs are carried in the blood, broken down or removed from the body. This study will look at the amount of drug in the blood and cells of the immune system for patients taking efavirenz, tenofovir and emtricitabine or atazanavir boosted with ritonavir, tenofovir and emtricitabine.

Participants: The population will comprise of 56 (6 for intensive PK and 50 for sparse sampling) HIV-infected adults currently adhering to an antiretroviral regimen containing efavirenz with tenofovir and emtricitabine and the same number and distribution of HIV-infected adults currently adhering to an antiretroviral regimen containing atazanavir boosted with ritonavir with tenofovir and emtricitabine.

Procedures (methods): This study will be completed at the University of North Carolina at Chapel Hill. There will be four groups of subjects: Efavirenz/tenofovir/emtricitabine Group A, Efavirenz/tenofovir/emtricitabine Group B, Atazanavir/ritonavir/tenofovir/emtricitabine Group A, and Atazanavir/ritonavir/tenofovir/emtricitabine Group B.

The initial six subjects (Group A) for intensive PK analysis for each regimen will be recruited from the the UNC ID Clinic or the Moses Cone Health System Infectious Diseases Clinic, and will be comprised of non-frail subjects not currently receiving interacting drugs. If subjects provide informed consent, timed blood samples will be obtained to determine pharmacokinetic parameters around an observed dose of one of the two study regimens. A whole blood sample will also be collected and stored for potential drug metabolizing enzymes and transporters genotyping in the future. Group A subjects will complete a follow-up visit after their sampling visit.

50 subsequent subjects (Group B) for each regimen will be screened simultaneously, with no more than 10 subjects enrolled for each regimen in Group B prior to the completion and analysis of Group A. These subjects will also be recruited from either site. Group B subjects will have one or two sampling visits with 1 to 4 blood samples obtained at each visit, with a stored sample for future genotyping obtained on one of the visits. Samples will be collected just prior to a dose, at 2 hours, between 4 and 6 hrs, and between 10 and 14 hours after a medication dose. These visits may coincide with the subjects' regularly scheduled visit to the clinic, or be scheduled separately, depending on the preference and availability of the subject.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patients
* Able to provide written informed consent
* Able to comply with their treatment regimen and study procedures
* Currently receiving either efavirenz/tenofovir/emtricitabine or atazanavir/ritonavir/tenofovir/emtricitabine as treatment for their HIV infection. Subjects must have been on the regimen for at least 2 weeks
* All women of reproductive potential must have a negative urine pregnancy test
* If participating in sexual activity that could lead to pregnancy, study participant must use at least one reliable method of contraception.

Exclusion Criteria:

* Displaying the fraility phenotype (Group A only)
* Receiving an interacting medication
* Having missed >3 doses of study medication in the past 30 days
* Patients who will not likely remain on the study regimen during the course of study participation.
* Anemia (hemoglobin <10 g/dL)
* Abnormal screening laboratory findings
* Pregnancy
* Breastfeeding
* Any condition that may interfere with follow-up or the ability to take the study medication appropriately.
* Any clinically significant surgical alterations of the alimentary track, that in the opinion of the investigators, alters the absorption pharmacokinetics of the drugs of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV Positive patients on a stable regimen consisting of either efavirenz/tenofovir/emtricitabine or atazanavir boosted with ritonavir/tenofovir/emtricitabine
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Clearance estimates for each drug, adjusted for age and frailty | From 0, 2, 4-6, and 10-14 hr post-dose blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Julie B Dumond, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Dumond JB, Francis O, Cottrell M, Trezza C, Prince HM, Mollan K, Sykes C, Torrice C, White N, Malone S, Wang R, Van Dam C, Patterson KB, Hudgens MG, Sharpless NE, Forrest A. Tenofovir/emtricitabine metabolites and endogenous nucleotide exposures are associated with p16(INK4a) expression in subjects on combination therapy. Antivir Ther. 2016;21(5):441-5. doi: 10.3851/IMP3017. Epub 2016 Jan 5. PMID 26731175